CLINICAL TRIAL: NCT07001358
Title: The Rufaida Project: Towards a Better Understanding of a Gut-vagina Axis by Investigating the Effects of Ramadan Fasting on Gut and Vaginal Microbial Communities
Brief Title: The Rufaida Project: Researching the Impact of Ramadan Fasting on the Gut and Vaginal Microbiome
Acronym: Rufaida
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: BUN B3002024000242
Record Dates: First submitted 2025-03-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-02

CONDITIONS: Intermittent Fasting; Gut Microbiome; Vaginal Microbiome
Keywords: Vaginal microbiome; Gut microbiome; Intermittent fasting; Ramadan; Gut-vagina axis; Citizen science
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Vaginal swabs with human and microbial DNA Stool swabs with human and microbial DNA Stool dry samples with human and microbial DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women participating in Ramadan: Healthy volunteers that plan on intermittent fasting during the month of Ramadan 2025. No food or drink will be consumed from sunrise until sundown

SUMMARY:
The body's systems are deeply connected, but they are often studied separately. A recent large-scale citizen-science project on women's health, called Isala, discovered a group of gut-related bacteria present in the vaginal microbiome. This finding supports the idea that gut and vaginal bacteria interact closely, a connection known as the gut-vagina axis. However, it remains unclear whether changes in gut bacteria influence the vaginal microbiome.

This discovery led to an exploration of how diet affects both the gut and vaginal microbiomes. In the gut, bacteria rely on carbohydrates from food, while in the vagina, bacteria feed on glycogen, a sugar stored in the vaginal lining. This glycogen is broken down into smaller sugars, which beneficial Lactobacillus bacteria use for fermentation. Since starch is a major source of these sugars, researchers suspect that a starch-rich diet may support Lactobacillus growth, which in turn promotes vaginal health.

To test this hypothesis, the Rufaida Project was launched. Ramadan is characterised by a fasting period of approximately one month during which participants abstain from eating between sunrise and sunset. Ramadan provides a unique opportunity to study how fasting affects the microbiome under controlled conditions.

In this study, 50 Muslim women will be asked to provide vaginal and stool samples at eight predetermined time points-before, during, and after Ramadan. These samples will be analysed using 16S rRNA amplicon sequencing to determine bacterial composition. Comparative analysis will be conducted between samples across different time points and anatomical sites. The objective is to understand how fasting and dietary changes influence the gut and vaginal microbiomes, and whether gut bacteria play a role in shaping vaginal health. Additionally, participants will complete weekly health questionnaires. An additional study group of up to 300 Muslim women will complete weekly questionnaires without providing biological samples.

This research could improve understanding of the links between diet, gut health, and vaginal health, potentially leading to new strategies for enhancing women's well-being through nutrition.

DETAILED DESCRIPTION:
The objective of this observational study is to examine the impact of fasting on the vaginal and gut microbiomes. The study population comprises healthy female volunteers of reproductive age who participate in Ramadan 2025. Participants will be enrolled in one of two study groups based upon their own selection.

Group One will include up to 50 women that provide vaginal and stool samples over a period of eight weeks: two weeks prior to Ramadan, throughout the four weeks of Ramadan, and two weeks following Ramadan. Sampling kits will be accompanied by an instruction brochure detailing standardized procedures to ensure reliable and consistent sample collection. In addition, participants in this group will complete a weekly questionnaire assessing general, mental, vaginal, gut, sexual, and reproductive health.

Group Two will consist of 300 women that complete the same weekly health questionnaire but will not provide biological samples.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older on the moment of registration
* Female (biological gender)
* Currently living in Belgium
* Sufficient knowledge of the Dutch language
* Participating in Ramadan
* Has signed the informed consent

Exclusion Criteria:

* Breastfeeding at the start of and during the study
* Current diagnosis of cancer and/or immunosuppressive therapy in the six months before the study
* Cardiovascular and metabolic conditions (such as diabetes, irritable bowel syndrome, etc.)
* Clinically significant tendency to bleed throughout history;
* Clinically significant abnormalities of the reproductive organs;
* Any other medical condition that, in the judgment of the principal investigator, warrants exclusion from the study;
* Use of oral/vaginal antibiotics/antimycotics in the 2 months prior to the study;
* Use of oral/vaginal pre-, pro-, and postbiotics (i.e., supplements in addition to diet) in the 2 weeks before and during the study;
* Ketogenic diet in the 2 weeks before and during the study;
* Vaginal douching during the study;
* Concurrent participation in another clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers participating in Ramadan 2025 will be recruited through various channels. The selected women can join select to join group 1 (n=50) that take biological samples and fill out weekly questionnaires, or group 2 (n=300) that fill out weekly questionnaires.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Characterizing the gut and vaginal microbiome in relation to dietary components and meal frequency during ramadan using 16S rRNA sequencing | up to 4 years
  To investigate the potential influence of dietary components and meal frequency on the gut and vaginal microbiome, vaginal and stool samples will be collected from participants before, during, and after a period of intermittent fasting (Ramadan). Bacterial community composition will be determined using 16S rRNA amplicon sequencing by Illumina MiSeq analysis. Bioinformatic tools will be employed to assess taxonomic profiles across different time points and anatomical sites. Particular attention will be given to correlations between gut- and vaginal-associated microbial taxa, with the aim of identifying bacterial signatures potentially shaped by dietary changes and fasting patterns. The analysis will further explore whether specific gut microbiota are associated with the presence or modulation of vaginal microbial communities, with a focus on health-promoting taxa such as Lactobacillus species.

SECONDARY OUTCOMES:
Determining changes in psychological well-being during Ramadan through longitudinal questionnaires | Up to 4 years
  Participants will complete comprehensive questionnaires at eight predetermined time points before, during, and after Ramadan. These questionnaires are designed to evaluate various aspects of mental health and social connectedness, including feelings of togetherness with family, community, and the surrounding environment. The researchers will specifically focus on the temporal changes in psychological well-being and social cohesion associated with the fasting period.
Characterization of metabolite profiles in vaginal and stool samples before, during, and after Ramadan fasting | Up to 4 years
  This study involves longitudinal analysis of vaginal and stool samples collected at baseline, during, and after a period of intermittent fasting (Ramadan). Metabolomic profiling will be performed to identify and quantify bacterial metabolites, with particular focus on changes associated with dietary modifications during fasting. Comparative analyses between vaginal and gut samples will be conducted to investigate potential correlations between microbial communities and their metabolic outputs across anatomical sites. Additionally, the research will emphasize the role of health-promoting microorganisms, including Lactobacillus and Saccharomyces species, in shaping the metabolite landscape.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Lebeer, Professor, Principal Investigator — Universiteit Antwerpen
Locations (1):
- University of Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The metadata of participants in the study will be made available in a restricted access repository.
  * For samples and data sharing, the researchers will work with the legal department to establish Material/Data Transfer Agreements.
  * Sequencing data are available at the European Nucleotide Archive.
  * Physical samples are their origin will be stored at the decentral hub of the Antwerp biobank.
  * Concerning non-identifiable sample meta-data that the researchers will use in analysis and will later be published will be put available with access control via the European Genome-Phenome Archive (EGA), where data can be accessed as described upon agreeing to the harmonized Data Access Agreement (developed by the European Union standards for in silico models for personalized medicine EU-STANDS4PM, https://doi.org/10.6084/m9.figshare.23904300).
Supporting Information: Study Protocol, ICF
Time Frame: Following publication, the results associated with each study will also be deposited in the Dryad repository, where they will be preserved indefinitely. Sequences will be stored to ENA (public databases) and NCBI. All samples will be registered in the Biobank using the SLIMS system.
Access Criteria: A guide to data access on the EGA is available at https://ega-archive.org/access/data-access, and a data access request will be processed within 2-3 months, pending evaluation by the data access committee (existing of lab members involved in the study), and processing by the EGA.

REFERENCES:
- See also: Webpage about the study for participants — https://isala.be/en/study/rufaida-en/
- See also: Blogpost explaining the study and studygroups to possible participants — https://isala.be/isala-zoekt-opnieuw-ramadan-deelneemsters/

DOCUMENTS (2):
  • Study Protocol (2025-02-13): https://cdn.clinicaltrials.gov/large-docs/58/NCT07001358/Prot_000.pdf
  • Informed Consent Form (2025-01-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT07001358/ICF_001.pdf